CLINICAL TRIAL: NCT01143311
Title: Role of microRNA in the Development of Cutaneous Squamous Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: CAILLON Cynthia, DRCI du CHU de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-PP-05
Record Dates: First submitted 2010-04-19; First posted 2010-06-14 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-06

CONDITIONS: Cancer of the Skin
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARM A (Other): 4 distinct biopsies will be taken
  1. in a non UV-exposed area (inner arm)
  2. in a UV-exposed area (external surface of the forearm)
  3. in a pretumoral region (actinic keratosis)
  4. inside the tumor
  Interventions: Genetic: Arm A

INTERVENTIONS:
Genetic: Arm A — 4 distinct biopsies will be taken
  1. in a non UV-exposed area (inner arm)
  2. in a UV-exposed area (external surface of the forearm)
  3. in a pretumoral region (actinic keratosis)
  4. inside the tumor

SUMMARY:
The aim of this study is to analyze the differential expression of the miR transcriptome in the distinctive stages of the development of cutaneous squamous cell carcinoma (C-SCC). In this aim the investigators plan to recruit a cohort of 20 patients suffering of C-SCC and to collect from each of them, biopsies corresponding to i) non UV-exposed areas ii) UV-exposed areas, iii) actinic keratosis and iv) tumoral regions. Total RNAs will be prepared from each biopsy and the miRNA profiles will be characterized using a dedicated miR array.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 40th, suffering of a C-SCC
* letter of consent signed by the patient
* to be registered to social security

Exclusion Criteria:

* Pregnant women or breastfeeding.
* Small C-SCC (size < 6mm)
* Allergy to Xylocaine
* All vulnerable (minor, adult guardianship…)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
miRNAs | 1 year
  We will select the miRNAs differently expressed between biopsies obtained respectively from areas of normal, pretumoral and tumoral areas (candidate miRs = miRs potentially involved in tumor transformation of epidermal keratinocytes). This will be assessed by analyzing in each of the biopsies from each patient, the expression of different miRs that are known to date, using a dedicated microarray, then by checking the data obtained by quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France